CLINICAL TRIAL: NCT01081574
Title: A Multicentre, International, Adaptive, Open-label, Repeated Administration Pharmacokinetic Study of Bilastine in Children From 2 to <12 Years of Age With Allergic Rhinoconjunctivitis or Chronic Urticaria
Brief Title: Pharmacokinetic Study of Bilastine in Children From 2 to < 12 Years of Age With Either Allergic Rhinoconjunctivitis (AR) or Chronic Urticaria (CU)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BILA 3009/PED; 2009-012013-22 (EudraCT Number)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Allergic Rhinoconjunctivitis; Chronic Urticaria
Keywords: Allergic Rhinitis; Seasonal Allergic Rhinitis; Perennial Allergic Rhinitis; Urticaria; Chronic Idiopathic Urticaria; Allergy; Sneezing; Nasal Itching; Rhinorrhea; Nasal Congestion; Wheals; Hives; Skin itching; Flare; Erythema
MeSH Terms: conditions — Chronic Urticaria; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial; Urticaria; Hypersensitivity; Sneezing; Rhinorrhea; Nasal Obstruction; Pruritus; Erythema | interventions — bilastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 10 mg Bilastine once daily for 7 days (Experimental): 10 mg Bilastine dispersible oral tablet
  Interventions: Drug: Bilastine

INTERVENTIONS:
Drug: Bilastine — 10 mg/qd/ 7 days.Oral dispersible tablets
  Other Names: Bilaxten

SUMMARY:
The conduct of this clinical trial is aimed at determining the most suitable dose regimen for children in different age groups, and secondarily to assess the safety and tolerability of bilastine in this paediatric population subset.

DETAILED DESCRIPTION:
The objective of this study is to assess the pharmacokinetics of bilastine in children (aged 2 to <12 years) with allergic rhinoconjunctivitis (seasonal allergic rhinitis [SAR] and/or perennial allergic rhinitis [PAR]) or chronic urticaria (CU) in order to ascertain that the systemic exposure attained with a dose of 10 mg/QD or lower is comparable to that achieved in adults and adolescents administered with a dose of 20 mg/QD.

Additional objectives are to describe the safety and tolerability of a repeated administration of bilastine in children with AR or CU.

ELIGIBILITY:
Inclusion Criteria:

1. Either sex aged from ≥ 2 to < 12 years of age. Female subjects must not be of child bearing potential.
2. Height and weight within a majority range (e.g., 25th through 75th percentile) of the subject's age and sex as provided in national tables.
3. Documented history of SAR/PAR or CU at the time of inclusion. Subjects must be symptomatic at screening as judged by the investigator.
4. A documented positive skin prick test or IgE test (RAST) for at least one seasonal or perennial allergen in children with AR obtained within the 12 months prior to inclusion.
5. Excepting AR or CU, judged to be in general good health based on medical history, physical examination and clinical laboratory tests, with a QTc duration on the ECG recorded at screening within the normal range (≤ 440 msec).
6. Written informed consent signed by the legal representative of the minor (his/her parent(s) or a person legally appointed if different from parent(s)) and, where applicable, assent signed by the child, according to local regulations.

Exclusion Criteria:

1. Female subjects of childbearing potential. If menarche occurs after study enrolment and during the dosing period, the subject should be discontinued from the treatment and followed up for safety as per protocol. Occurrence of menarche in the course of the study should always be documented.
2. Intake of another investigational medication in another clinical study within 30 days prior to the first study drug intake.
3. Clinically significant ECG abnormalities as judged by the investigator (e.g., Wolff-Parkinson-White [WPW] syndrome, long QT syndrome).
4. Known allergy/hypersensitivity to the study drug or its inactive ingredients.
5. Any clinical conditions or circumstances that in the opinion of the investigator would make the subject unsuitable for the study (e.g., hepatic impairment, renal impairment, mental impairment, cardiac disease).
6. Subjects with known positive Hepatitis B surface antigen (Hbs Ag), or Hepatitis C antibody or who are known to be human immunodeficiency virus (HIV) positive. No testing will be required for this study.
7. Subjects who are expected to take during the study period or have taken any of the following medications prior to inclusion in the study and have not complied with the specified wash out period of 7 days unless otherwise noted:

   * Oral corticosteroids.
   * Oral antihistamines: loratadine, desloratadine, and fexofenadine.
   * Anti-leukotrienes
   * Amoxicillin, benzylpenicillin, and macrolide antibiotics and imidazolic antifungals (systemic)
   * Omeprazol
   * Aspirin, ibuprofen
   * Carbamazepine
   * St. John's Wort (15 days)
8. Hypersensitivity to H1 antihistamines or benzimidazoles.
9. Ingestion of citrus fruits and cranberries or any fruit juice or any other well known PgP or organic anion transporter polypeptide (OATP) inhibitor, inducer, or substrate (see Appendix C) within 7 days prior to first dose of study medication.
10. Mentally disabled minors or Minors who by official order have been institutionalised (e.g., in orphanages) must be excluded from participation.
11. Minors who explicitly refuse to take part in the study.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the pharmacokinetics of bilastine in children (aged 2 to <12 years) with allergic rhinoconjunctivitis (seasonal allergic rhinitis and/or perennial allergic rhinitis [SAR/PAR]) or chronic urticaria (CU) | 1 day (visit 3, Day 7)
  Determination of plasma concentrations versus time (between 1 and 6 samples per subject at various time intervals after dosing according to an optimised sampling protocol) in order to perform a population pharmacokinetic analysis.
  For Group A, samples of venous blood will be just prior to dose administration, and at 0.25, 0.5, 0.8, 1.0, 1.2, 1.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, and 24.0 hours after dose administration.
  For Group B samples of venous blood will be just prior to dose administration, and at 0.25, 0.5, 1.0, 1.5, 3.0, 6.0, 8.0, 10.0, and 12.0 hours after dose administration.

SECONDARY OUTCOMES:
The secondary objectives are to describe the safety and tolerability of a repeated administration of bilastine in the aforementioned paediatric subset with allergic rhinoconjunctivitis (SAR/PAR) or chronic urticaria (CU). | 5 weeks
  Safety will be assessed during the study by monitoring adverse events (AEs), clinical laboratory test results (urinalysis, blood chemistry, and haematology), vital signs (including blood pressure, respiration, temperature, and heart rate, supine and standing), electrocardiogram (ECG) results, and abnormal findings upon physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Wahn, Prof. Dr., Principal Investigator — International Coordinating Investigator. Charité - Universitätsmedizin Berlin (Germany); Regina Föster-Holst, Prof. Dr., Principal Investigator — Universitäts-Hautklinik Kiel (Germany); Belén Sádaba, Dr., Principal Investigator — Clínica Universitaria de Navarra (Spain); Gunilla Hedlin, Prof. Dr., Principal Investigator — Karolinska University Hospital; Stefan Zielen, Prof. Dr., Principal Investigator — J.W. Goethe-Universität Frankfurt (Germany); Lennart Nordvall, Prof. Dr, Principal Investigator — Children's Hospital at Uppsala University Hospital (Sweden); Peter Le Souef, Prof. Dr., Principal Investigator — Princess Margaret Hospital for Children (Australia); Noel E Cranswick, Prof. Dr., Principal Investigator — Royal Children's Hospital
Locations (7):
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Subiaco, Western Australia
- Germany (3):
  - Charité - Universitätsmedizin. Campus Virchow-Klinikum. Klinik für Pädiatrie mit Schwerpunkt Pneumologie/Immunologie, Berlin
  - Klinikum der Johann-Wolfgang-Goethe-Universität Frankfurt, Franfurt
  - Universitäts-Hautklinik, Kiel
- Sweden (2):
  - Karolinska University Hospital. Astrid Lindgren's Hospital, Stockholm
  - Children's Hospital at Uppsala University Hospital, Uppsala

REFERENCES:
- [Background] Jauregizar N, de la Fuente L, Lucero ML, Sologuren A, Leal N, Rodriguez M. Pharmacokinetic-pharmacodynamic modelling of the antihistaminic (H1) effect of bilastine. Clin Pharmacokinet. 2009;48(8):543-54. doi: 10.2165/11317180-000000000-00000. PMID 19705924
- [Background] Zuberbier T, Oanta A, Bogacka E, Medina I, Wesel F, Uhl P, Antepara I, Jauregui I, Valiente R; Bilastine International Working Group. Comparison of the efficacy and safety of bilastine 20 mg vs levocetirizine 5 mg for the treatment of chronic idiopathic urticaria: a multi-centre, double-blind, randomized, placebo-controlled study. Allergy. 2010 Apr;65(4):516-28. doi: 10.1111/j.1398-9995.2009.02217.x. Epub 2009 Oct 23. PMID 19860762
- [Background] Horak F, Zieglmayer P, Zieglmayer R, Lemell P. The effects of bilastine compared with cetirizine, fexofenadine, and placebo on allergen-induced nasal and ocular symptoms in patients exposed to aeroallergen in the Vienna Challenge Chamber. Inflamm Res. 2010 May;59(5):391-8. doi: 10.1007/s00011-009-0117-4. Epub 2009 Nov 27. PMID 19943178
- [Background] Kuna P, Bachert C, Nowacki Z, van Cauwenberge P, Agache I, Fouquert L, Roger A, Sologuren A, Valiente R; Bilastine International Working Group. Efficacy and safety of bilastine 20 mg compared with cetirizine 10 mg and placebo for the symptomatic treatment of seasonal allergic rhinitis: a randomized, double-blind, parallel-group study. Clin Exp Allergy. 2009 Sep;39(9):1338-47. doi: 10.1111/j.1365-2222.2009.03257.x. Epub 2009 May 4. PMID 19438584
- [Background] Bachert C, Kuna P, Sanquer F, Ivan P, Dimitrov V, Gorina MM, van de Heyning P, Loureiro A; Bilastine International Working Group. Comparison of the efficacy and safety of bilastine 20 mg vs desloratadine 5 mg in seasonal allergic rhinitis patients. Allergy. 2009 Jan;64(1):158-65. doi: 10.1111/j.1398-9995.2008.01813.x. PMID 19132976